CLINICAL TRIAL: NCT05072548
Title: Evaluating the Effectiveness of the ABCs of SLEEPING Mobile Applicable
Brief Title: The ABCs of SLEEPING: Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38732
Record Dates: First submitted 2021-07-28; First posted 2021-10-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Sleep Problems; Behavioural Insomnia of Childhood
Keywords: School aged children; Sleep problems; Behavioural insomnia; Smartphone intervention; Behavioural intervention
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Masking Description: Participants will be made aware what group they are randomized to (i.e., control or treatment group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive access to the ABCs of SLEEPING Intervention.
  Interventions: Behavioral: The ABCs of SLEEPING
- Control group (No Intervention): The control group arm does not receive the ABCs of SLEEPING intervention. This arm is free to access other resources while enrolled in the study. After the post-test follow up time point, the control group arm will be able to access the intervention.

INTERVENTIONS:
Behavioral: The ABCs of SLEEPING — The intervention is comprised of three components. The first is a sleep check-in which is a questionnaire that is evidence based and evaluates what areas of sleep parents can work on. The second component is the sleep report which summarizes to the parent what areas they're doing well in (i.e., within the ABCs of SLEEPING mnemonic described above) and what areas they can improve on. The third component of this intervention are the "sleep tips" which are sleep recommendations that are customized based on the identified areas of sleep the parents are suggested to work on.
  Arms: Intervention

SUMMARY:
This trial will examine the effectiveness of a mobile applicable intervention called the "ABCs of SLEEPING". This intervention provides parents with prioritized/customized sleep recommendations and a sleep report based on their responses to the "Sleep check-in". This app is evidence-based and developed by sleep researchers and its aim is to provide accessible evidence-based sleep information for parents of children aged 6 to 12 years of age.

DETAILED DESCRIPTION:
An evidence-based approach to treating sleep problems in school-aged children is to follow a stepped approach where interventions more easily implemented with fewer side effects (i.e., psychoeducation and implementing healthy sleep practices) are implemented first, followed by more involved approaches (i.e., behavioural intervention), and only using those with potential side effects as a final approach (i.e., medication). While there have been interventions developed for all of the above noted approaches, there are practical barriers (e.g., time and cost) as well as system barriers (e.g., healthcare professionals reporting a lack of training, knowledge, and time to provide evidence-based sleep care). Together, these barriers impact the ability of parents to access sleep intervention within this stepped approach. Given the high prevalence of internet use in North America, there is a growing trend for interventions to be adapted to online formats which addresses these accessibility barriers so that these interventions can reach most families with access to the internet. A smartphone app-based mode of intervention delivery is useful for accessibility and convenience reasons (e.g., no time cost for attending program/intervention sessions for busy parents, cost-effectiveness, etc.). Additionally, delivering sleep intervention via a smartphone app has the strong potential for effectiveness as they are delivered in a home setting (i.e., where new intervention practices are to occur). The investigator's research team has developed a smartphone app intervention called "ABCs of SLEEPING" which was initially developed to be a mnemonic to draw attention to the important factors that must be considered for healthy sleep practices for children: 1) age-appropriate bedtimes and wake-times with consistency, 2) schedules and routines, 3) location, 4) no electronics in the bedroom or before bed, 5) exercise and diet, 6) positivity, 7) independence when falling asleep, and 8) needs met during the day, 9) equal great sleep. The ABCs intervention includes three components. The first component is the ABCs of SLEEPING questionnaire that assesses the child's sleep practices using parent's responses to questions within each of the ABCs of SLEEPING healthy sleep practice areas. These responses algorithmically determine the feedback received on the second component, the sleep report card, which provides parents with feedback on each healthy sleep practice area. Feedback is provided based on a star system, with one star denoting the sleep practice area to be high priority (i.e., the healthy sleep practice recommendations are not being met), two stars denoting medium priority (i.e., the healthy sleep practice recommendations are not being fully met), and three stars denoting low priority (i.e., the healthy sleep practice recommendations are being fully met). The third component, the sleep tips, are then organized for the user in terms of priority. Priority is based on the star system described above, in combination with the robustness of the evidence for the healthy sleep recommendation. For example, if one star was received for both use of electronics at night and exercising prior to bed, use of electronics would be prioritized over exercising before bed based on the strength of the extant literature for this recommendation. To date, the ABCs of SLEEPING intervention has undergone evaluation in terms of its usability (i.e., usability, usefulness, desirability, etc.) and feasibility (i.e., acceptability, implementation, and preliminary efficacy). The next step in this research is to evaluate the ABCs of SLEEPING intervention for its effectiveness using increasing control (i.e., a control group and controlling for variables like sleep medication).

This effectiveness trial will be composed of three study periods. The first period is the "pre-test" period where baseline measures of the Children's Sleep Habits Questionnaire, Pediatric Insomnia Severity Index, Bedtime Routines Questionnaire, Actigraph/Sleep Diary, as well as demographics (i.e., measured using a Demographics Questionnaire) are collected. Following this pre-test period, parents will be randomized to either to the treatment or the control group. Parents randomized to the treatment group will receive the ABCs of SLEEPING intervention for a 4-week period. Parents in the intervention group will no longer have access to the intervention after this 4-week period concludes. Parents in the control group are not required to complete any study measures during this time period. Following this "intervention period" is the "post-test" period. During the post-test period, parents will complete again the study's measures (i.e., The Children's Sleep Habits Questionnaire, Pediatric Insomnia Severity Index, Bedtime Routines Questionnaire, and Actigraph/Sleep Diary). After completing the post-test period, the study will conclude. Additionally, parents in the control group will receive the intervention for a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Canada
* Have internet/computer and smartphone access and an email account for the completion of online questionnaire and for accessing the intervention
* Be comfortable reading and writing in English
* child has at least 1 behaviourally-based sleep problem (i.e., either difficulty falling asleep, staying asleep, and early morning awakenings)

Exclusion Criteria:

* Child should not have a significant mental or physical health condition (i.e., defined as the child being ambulatory, not hospitalized or in residential care, and able to complete developmentally appropriate daily activities as expected for their age)
* Child should not have a known intrinsic sleep disorder (e.g., sleep apnea)
* Child should not be taking a sleep medication

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Children's Sleep Habits Questionnaire (i.e., child sleep habits measure) | Measured once at pre-test and once at post-test (i.e., 6-week follow up) to examine change in sleep habits.
  This questionnaire was designed as a sleep screening instrument for school-aged children that yields final scores across eight subscales: bedtime resistance, sleep resistance, parasomnia, sleep disordered breathing, night-wakings, daytime sleepiness, sleep anxiety, and sleep onset delay, as well as a summative score, called the Total Sleep Disturbance score. This is the investigator's primary outcome measure because the ABCs of SLEEPING is aimed at improving children's sleep habits.

SECONDARY OUTCOMES:
Pediatric Insomnia Severity Index (i.e., pediatric insomnia severity measure) | Measured once at pre-test and once at post-test (i.e., 6-week follow up) to examine change in pediatric insomnia severity.
  The Pediatric Insomnia Severity Index assesses sleep onset problems using parental report of sleep maintenance problems, daytime sleepiness, and nocturnal sleep duration. This questionnaire will be used to describe the severity of insomnia in this sample, as well as to assess change in insomnia severity.
Actigraphy (i.e., sleep onset latency measure). | Measured for 5-7 days at pre-test, and 5-7 days at post-test (i.e., 6-week follow up) to examine change in sleep onset latency (i.e., objective measures of sleep).
  An actigraph is a battery-operated, watch-like device, most often worn on the non-dominant wrist, that collects movement information using accelerometer technology. Previous studies have shown that the commercial software algorithms used to analyze actigraphy data provide valid and reliable estimates of when participants are asleep and awake, as well as a means of assessing sleep quality variables such as sleep latency and duration. For the current study, Philips actigraphs will be used. The participant's child will wear an actigraph for the purposes of collecting objective information about sleep onset latency (how quickly the child falls asleep). Note that actigraphy is used for measuring both sleep onset latency and sleep efficiency. The investigators have described these as two separate outcome measures that are measured using the same tool (i.e., actigraphy).
Sleep Diary | Measured for 5-7 days at pre-test, and 5-7 days at post-test (i.e., 6-week follow up) to examine change in sleep onset latency and sleep efficiency (i.e., the sleep diary is used alongside actigraphy data as an objective measure of sleep).
  This study will utilize a brief 8-item sleep diary to collect parent-reported sleep variables (e.g., "what time was your child down for the night?"). This questionnaire will be utilized to help score actigraphy data by examining corresponding information.
Actigraphy (i.e., sleep efficiency measure). | Measured for 5-7 days at pre-test, and 5-7 days at post-test (i.e., 6-week follow up) to examine change in sleep efficiency (i.e., objective measures of sleep).
  An actigraph is a battery-operated, watch-like device, most often worn on the non-dominant wrist, that collects movement information using accelerometer technology. Previous studies have shown that the commercial software algorithms used to analyze actigraphy data provide valid and reliable estimates of when participants are asleep and awake, as well as a means of assessing sleep quality variables such as sleep latency and duration. For the current study, Philips actigraphs will be used. The participant's child will wear an actigraph for the purposes of collecting objective information about sleep efficiency (the percentage of time scored as asleep during the sleep period from the time the child goes to bed to the time the child gets out of bed in the morning). Note that actigraphy is used for measuring both sleep onset latency and sleep efficiency. The investigators have described these as two separate outcome measures that are measured using the same tool (i.e., actigraphy).

CONTACTS AND LOCATIONS:
Overall Officials: Penny Corkum, PhD, Principal Investigator — IWK Health Centre; Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This trial will be reported at a group level only, not individual participant level.